CLINICAL TRIAL: NCT02714439
Title: Low-Cost Imaging for Cervical Cancer Prevention in the Texas Lower Rio Grande Valley
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI has left the institution
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: M.D. Anderson Cancer Center (Other); The University of Texas Health Science Center, Houston (Other); William Marsh Rice University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0014-0302; NCI-2016-00729 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-03-16; First posted 2016-03-21 (Estimated); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Malignant Neoplasms of Female Genital Organs
Keywords: Malignant neoplasms of female genital organs; Cervical Cancer Prevention; Abnormal Pap test; Positive HPV test; History of cervical dysplasia; Colposcopy; Proflavine; Proflavine hemisulfate; High-Resolution Microendoscopy; HRME; Human papillomavirus
MeSH Terms: interventions — Proflavine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- High-Resolution Microendoscopy (HRME) (Experimental): After standard colposcopy examination performed, participants undergo a high-resolution microendoscopy imaging procedure. Proflavine 0.01% is applied to the cervix, then high-resolution microendoscopy imaging procedure performed. Standard colposcopy procedure will then continue.
  Interventions: Drug: Proflavine; Procedure: High-Resolution Microendoscopy (HRME)

INTERVENTIONS:
Drug: Proflavine — Proflavine 0.01% applied to the cervix before high-resolution microendoscopy imaging procedure performed.
  Other Names: Proflavine hemisulfate
Procedure: High-Resolution Microendoscopy (HRME) — High-resolution microendoscopy imaging procedure performed after colposcopy exam. Standard colposcopy procedure will then continue. Entire HRME imaging procedure should add less than 10 minutes to the standard colposcopy exam.

SUMMARY:
The purpose of this study is to evaluate a different type of medical equipment called "High-Resolution Microendoscope" (HRME) for the diagnosis of cervical pre-cancerous lesions and cervical cancer. The investigators want to compare patients' clinical findings using the current equipment used in clinic with the clinical findings using new equipment we are testing on this research project. If the new equipment is proven to give comparable findings with current equipment being used, doctors might be able to offer a diagnosis and treat cervical lesions in one visit. It might not be necessary to wait for cervical biopsies to come back before women would receive the indicated treatment. Study subjects are being asked to participate because they have been diagnosed with an abnormal Papanicolaou (Pap) PAP smear, positive human papillomavirus (HPV) test or history of cervical dysplasia and need to have a colposcopic examination to determine the reason for abnormal results and receive treatment.

DETAILED DESCRIPTION:
Investigators will start the participants' examination with colposcopic evaluation using current equipment as determined by standard of care. But, if cervical biopsies are indicated, before performing biopsies, for research purposes only - investigators will:

* Apply a substance called Proflavine 0.01% to participants' cervix
* Investigators will re-evaluate participants' cervix with the new equipment being tested:The High- Resolution Microendoscope
* After completing this re-evaluation, investigators will continue with the standard of care protocol and will perform participants' cervical biopsies if indicated.

The entire re-evaluation with the new equipment should add less than 10 minutes to the standard examination.

When a woman is found to have an abnormal PAP smear, depending on the findings and clinical history, most women will need to be further evaluated with a colposcope in order to understand the reason for the abnormal PAP and determine the best treatment. This is called colposcopic examination and it is the standard of care. This procedure is performed in the clinic, patient is positioned on the examining table the same way she is positioned for a Papanicolaou (Pap) smear, a speculum is placed inside the vaginal canal, and certain substances are applied to the cervix in order to identify cervical lesions. These substances might include acetic acid and/or Lugol's iodine solution. The application of these substances helps to delineate the abnormal cervical areas that might need to be biopsied. For the purpose of this research study, before obtaining the biopsies, a second evaluation will be performed using the equipment that is being studied (High- Resolution Microendoscope) and using a different substance that will be applied to the cervix. This substance is called Proflavine 0.01%. . This second evaluation should not take more than 10 minutes. After completing this second evaluation, participants' clinical examination and clinical visit should continue as routine.

The anticipated total number of subjects involved in the study will be 150 women. All these anticipated participating women would be from The University of Texas Medical Branch (UTMB), Su Clinica and UT Health Science Center (UT-HSC) Mobile Van. The length of time for participation is 1 year. However, during the participants' year of enrollment she might have only one examination, during one of her visits,using the research equipment.

ELIGIBILITY:
Inclusion Criteria:

1. Women with an abnormal Pap test, positive HPV test or any history of cervical dysplasia
2. Women with an intact cervix (patients who have undergone previous LEEP, cone and/or cryotherapy are eligible)
3. Women of childbearing potential must have a negative urine or serum pregnancy test
4. Women who are at least 21 years of age or older
5. Ability to understand and the willingness to provide informed consent and sign a written Informed Consent Document (ICD)
6. For patients that present to clinic to have a cervical excisional procedure (LEEP) for an already confirmed diagnosis of high grade cervical dysplasia, HRME imaging study will be performed and cervical biopsies might be taken for research purposes only. Since these patients have already the confirmed diagnosis of high-grade cervical dysplasia, any extra biopsies taken will be for research purposes only and our research fund will pay them

Exclusion Criteria:

1. Women < 21 years of age
2. Women who have undergone a hysterectomy with removal of the cervix
3. Women with a known allergy to proflavine, acriflavine, or iodine
4. Women who are pregnant or nursing
5. Patients unable or unwilling to provide informed consent or sign a written Informed Consent Document (ICD)

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of the High-Resolution Microendoscopy (HRME) | 1 day
  Successful outcome defined as concordance between the diagnosis using HRME imaging and the most severe histologic diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Rodriguez, MD, Principal Investigator — University of Texas Medical Branch (UTMB); Kathleen Schmeler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas Medical Branch Cancer Stop McAllen Clinic, McAllen, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Texas Medical Branch web site — http://www.utmb.edu